CLINICAL TRIAL: NCT06617416
Title: A Randomized, Double-blind, Multicenter Phase III Study to Evaluate the Consolidation Therapy of AK104 Versus Sugemalimab in Patients With Unresectable Locally Advanced Non-Small Cell Lung Cancer Who Have Not Progressed After Concurrent or Sequential Chemoradiotherapy
Brief Title: A Study of AK104 in Subjects With Unresectable Locally Advanced NSCLC
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Akeso (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AK104-309
Record Dates: First submitted 2024-09-25; First posted 2024-09-27 (Actual); Last update posted 2025-03-12 (Actual); Status verified 2025-03

CONDITIONS: NSCLC (Non-small Cell Lung Cancer)
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — sugemalimab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- AK104 group (Experimental): AK104 Q3W
  Interventions: Drug: Cadonilimab (AK104)
- Sugemalimab group (Active Comparator): Sugemalimab 1200mg Q3W
  Interventions: Drug: Sugemalimab

INTERVENTIONS:
Drug: Cadonilimab (AK104) — AK104 ivgtt Q3W
  Arms: AK104 group
Drug: Sugemalimab — 1200mg Q3W
  Arms: Sugemalimab group

SUMMARY:
This study compares the efficacy and safety of AK104 versus Sugemalimab as consolidation therapy in patients with unresectable, locally advanced NSCLC who have not progressed following concurrent or sequential chemoradiotherapy.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects must sign the written informed consent form (ICF) voluntarily.
2. Age ≥18 years.
3. Histologically or cytologically confirmed unresectable locally advanced (Stage III) NSCLC.
4. Absence of known EGFR sensitive mutations and negative for ALK and ROS1 fusions.
5. Concurrent or sequential chemoradiotherapy completed 1 to 42 days prior to the first dose.
6. Chemotherapy regimens should be in accordance with current clinical guidelines.
7. Consolidation chemotherapy is not allowed after radiotherapy.
8. Total dose of radiotherapy is 60Gy±10% (54Gy-66Gy).
9. No disease progression after concurrent or sequential chemoradiotherapy.
10. ECOG performance status score of 0-1.
11. Expected survival of over 3 months.
12. Adequate organ and bone marrow function.

Exclusion Criteria:

1. The histopathology contains any component of small cell lung cancer.
2. Currently participating in another interventional clinical study.
3. Previously received immunotherapy, biotherapy, anti-angiogenic drugs, or small molecule targeted drugs.
4. Patients with clinically significant cardio-cerebrovascular or venous thromboembolic diseases.
5. Prior malignancy active within the previous 3 years except for the locally curable cancers that have been apparently cured.
6. Tumor invades important vessels or organs.
7. Experienced acute exacerbation of chronic obstructive pulmonary disease or asthma within 4 weeks prior to the first dose.
8. Presence of interstitial lung disease that requires treatment.
9. Toxicities of prior anticancer therapy have not resolved to ≤ Grade 1 (NCI-CTCAE version 5.0).
10. Experienced severe infection within 4 weeks prior to the first dose.
11. Underwent major surgery or experienced severe trauma within 4 weeks prior to the first dose.
12. Any condition that required systemic treatment with corticosteroids (> 10 mg daily prednisone or equivalent) or other immunosuppressive agents within 14 days prior to the first dose.
13. Active autoimmune diseases or history of autoimmune diseases that may relapse.
14. Previous history of severe hypersensitivity reactions to other monoclonal antibodies.
15. Previous organ transplantation or allogeneic hematopoietic stem cell transplantation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 560 (Estimated)
Dates: Start 2024-11-12 (Actual); Primary Completion 2026-10-28 (Estimated); Study Completion 2028-12-30 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival (PFS) assessed by INV | 3 years
  PFS is defined as the time from randomization until the first documentation of disease progression or death due to any cause, whichever occurs first (based on RECIST Version 1.1).

SECONDARY OUTCOMES:
OS | 5 years
  Time from randomization to death
6-month PFS rate assessed by INV | 3 years
  PFS rate at 6 months
AEs | 3 years
  Adverse events incidence and severity, clinically significant abnormal laboratory test results.

CONTACTS AND LOCATIONS:
Overall Officials: Jinming Yu, MD, Principal Investigator — Shandong Cancer Hospital and Institute
Locations (1):
- Cancer Hospital of Shandong First Medical University, Jinan, China

IPD SHARING:
Plan to Share IPD: No